CLINICAL TRIAL: NCT03446872
Title: Post Marketing Surveillance Study for ONIVYDE® in South Korea
Status: Completed | Type: Observational
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Other Study IDs: 331602
Record Dates: First submitted 2018-02-12; First posted 2018-02-27 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — irinotecan sucrosofate; Fluorouracil; Leucovorin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- All Study Participants: Patients in South Korea with a diagnosis of metastatic pancreatic cancer who have been prescribed ONIVYDE
  Interventions: Drug: ONIVYDE; Drug: 5-fluorouracil; Drug: Leucovorin

INTERVENTIONS:
Drug: ONIVYDE — irinotecan liposome injection
Drug: 5-fluorouracil — a nucleoside metabolic inhibitor
  Other Names: 5-FU; fluorouracil
Drug: Leucovorin — an active metabolite of folic acid
  Other Names: LV

SUMMARY:
The purpose of this study is to characterize the safety of ONIVYDE when used under standard clinical practice in South Korea; and to describe effectiveness in patients receiving ONIVYDE in combination with 5-fluorouracil (5-FU) and leucovorin for the treatment of metastatic pancreatic cancer under standard clinical care in South Korea.

ELIGIBILITY:
Inclusion Criteria:

Patients who are prescribed ONIVYDE per investigator's judgment shall be included if:

* Patient / legally authorized representative/ family member gave written informed consent
* Patient is indicated for treatment according to ONIVYDE South Korea prescribing information
* Histologically or cytologically confirmed adenocarcinoma of exocrine pancreas
* Documented metastatic disease
* Patient deemed not eligible or failed previous treatment with gemcitabine or gemcitabine containing therapy
* Adequate hepatic, renal and hematological function

Exclusion Criteria:

* Patients enrolled in Servier sponsored ONIVYDE Registry or any other Servier sponsored ONIVYDE study
* Patients who have experienced severe hypersensitivity reaction to ONIVYDE or Irinotecan HCL
* Patients with new or progressive dyspnea, cough, and fever, pending diagnostic evaluation of interstitial lung disease. Patients with confirmed diagnosis of interstitial lung disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in South Korea with a diagnosis of metastatic pancreatic cancer.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2020-08-29 (Actual); Study Completion 2020-08-29 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs) | Throughout the study period approximately 4 years
  Number of AEs by seriousness and severity
Grade 3 and 4 neutropenia cases | Throughout the study period approximately 4 years
  Frequency of Grade 3 and 4 neutropenia cases

SECONDARY OUTCOMES:
Visit Information: Number of Visit Types | Throughout the study period approximately 4 years
  Number of: Outpatient/office Visits, In-hospital Visits, Phone Visits, or Other Types Visits
Visit Information: Reason for Visits | Throughout the study period approximately 4 years
  Number of: Scheduled Visits, Emergency Visits, Other Types Visits
Median Dose of ONIVYDE | Throughout the study period approximately 4 years
  Median Dose of ONIVYDE administered during the study period
Median Dose of fluorouracil | Throughout the study period approximately 4 years
  Median Dose of fluorouracil administered during the study period
Median Dose of Leucovorin | Throughout the study period approximately 4 years
  Median Dose of Leucovorin administered during the study period
Overall response | Throughout the study period approximately 4 years
  Response duration usually is measured from the time of initial response until documented tumor progression.
Overall Survival | Throughout the study period approximately 4 years
  The time from enrollment to death from any cause, is a direct measure of clinical benefit to a patient.
Progression free survival | Throughout the study period approximately 4 years
  The time elapsed between treatment initiation and tumor progression or death from any cause.
Quality of Life assessment (EQ-5D-5 L Health Questionnaire) | Baseline, and then every 3 weeks, and at the end of study visit up to approximately 4 years
  The instrument that measures conceptual domains of quality of patients' well-being.

CONTACTS AND LOCATIONS:
Locations (10):
- South Korea (10):
  - Konyang University Hospital, Daejeon
  - National Cancer Center, Gyeonggi-do
  - Severance Hospital, Yonsei University Health System - Gastroenterology, Seoul
  - Severance Hospital, Yonsei University Health System - Oncology, Seoul
  - ASAN Medical Center, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center - Oncology, Seoul
  - The Catholic University of Korea Seoul St.Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Ajou University Hospital, Suwon

IPD SHARING:
Plan to Share IPD: No